CLINICAL TRIAL: NCT04497571
Title: Immediate Load in Dental Implants Using Conventional Drilling and Piezoelectric Osteotomy on Aesthetic Zone: Randomized Clinical Trials.
Brief Title: Immediate Load in Dental Implants Using Conventional Drilling and Piezoelectric Osteotomy on Aesthetic Zone.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Isabel Godoy Reina, Professor of Master of Periodontology and Implant Dentistry, PhD student., Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IGR UGranada
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Dental Implants; Tooth Loss
Keywords: Dental implants; Piezoelectric osteotomy; Piezoelectric surgery; Immediate load
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Intervention Model Description: Randomized clinical trials.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezoelectric osteotomy (Experimental): Implant placement by piezoelectric osteotomy
  Interventions: Procedure: Piezoelectric osteotomy.
- Conventional drilling (Active Comparator): Implant placement by conventional drilling
  Interventions: Procedure: Conventional drilling

INTERVENTIONS:
Procedure: Piezoelectric osteotomy. — Implants placed using the ultrasonic technique.
  Arms: Piezoelectric osteotomy
Procedure: Conventional drilling — Implants placed using drilling technique
  Arms: Conventional drilling

SUMMARY:
Compare the survival rate of the implants placed using the ultrasonic technique and placed using conventional drilling, with an immediate load on the aesthetic zone.

DETAILED DESCRIPTION:
Main goals.

Compare the survival rate of the implants placed using the ultrasonic technique and placed using conventional drilling, with an immediate load on the aesthetic zone.

Specific goals.

* Evaluate the marginal peri-implant bone loss after the healing period through radiographs, from the day of surgery, to a month, to 3 and 6 months after and a year after the implants insertion.
* Evaluate the primary stability of each individual implant the day of their insertion to verify their load on the moment of surgery and also compare the values of each preparation techniques of implant bone preparation.
* Evaluate the secondary stability of each individual implant and compare the values of each preparation techniques.
* Evaluate the peri-implant clinic parameters within 3 and 6 months and a year after the insertion of the implants through these variables: probing depth and bleeding of probing.

ELIGIBILITY:
Inclusion Criteria:

* Absence of teeth on the aesthetic zone, whether its an incisor, canine or premolar.
* 3 months after the dental extraction without alveolar scar tissue remains.
* Bone availability of at least 5mm of width and 13mm of length.
* At least 2 to 3 mm of soft tissue for the establishment of an adequate peri-implant biological width.
* Oclusal pattern that ensures prosthetic success.
* Implants need to have at least a 35 N and 70 ISQ index to be loaded.
* Index of plaque < 20% and/or inactive periodontal disease.

Exclusion Criteria:

* Acute myocardial infarction in the last 2 months.
* Uncontrolled coagulation disorders
* Uncontrolled diabetes (HbA1c> 7.5%).
* Radiotherapy on head/neck in the last 24 months.
* Immunocompromised patient.
* History of medication related to osteonecrosis of the jaws.
* Psychiatric disorders, alcohol, drugs and large smokers (>10 cigarrillos).
* Plaque index > 20%.
* Need for simultaneous or previous peri-implant guided bone regeneration procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Loss | 1 month
  To compare MBL measured using radiographs.
Marginal Bone Loss | 3 months
  To compare MBL measured using radiographs.
Marginal Bone Loss | 6 months
  To compare MBL measured using radiographs.
Marginal Bone Loss | 12 months
  To compare MBL measured using radiographs.

SECONDARY OUTCOMES:
Primary stability | Baseline
  Implant Stability Quotient Values (Osstell ISQ, Osstell USA) obtained from implants in study site, recording immediately.
Secondary stability | 3 months
  Implant Stability Quotient Values (Osstell ISQ, Osstell USA) obtained from implants in study site, recording at 3 months.
Probing depth | 3,6,12 months
  Evaluate the peri-implant clinic parameters within 3 and 6 months and a year after the insertion of the implants through these variables: probing depth and bleeding of probing.
Bleeding of probing | 3,6,12 months
  Evaluate the peri-implant clinic parameters within 3 and 6 months and a year after the insertion of the implants through these variables: probing depth and bleeding of probing.
Survival rate | 3,6,12 months
  To measure implant success rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Isabel Godoy Reina, Almería, Spain

IPD SHARING:
Plan to Share IPD: Undecided